CLINICAL TRIAL: NCT02606903
Title: Randomized, Single-dose, Parallel-arm, Open-label Phase I Trial to Investigate and Compare the Pharmacokinetics, Safety and Tolerability of BI 695501 Administered Subcutaneously Via Prefilled Syringe or Autoinjector
Brief Title: Pharmacokinetics and Safety of BI 695501 Administered Via Prefilled Syringe or Autoinjector
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1297.6; 2015-003029-32 (EudraCT Number)
Record Dates: First submitted 2015-11-16; First posted 2015-11-17 (Estimated); Results first posted 2018-12-27 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-06

CONDITIONS: Healthy

ARMS (2):
- BI 695501 prefilled syringe (Experimental)
  Interventions: Drug: BI 695501 prefilled syringe
- BI 695501 autoinjector (Experimental)
  Interventions: Drug: BI 695501 autoinjector

INTERVENTIONS:
Drug: BI 695501 prefilled syringe
  Arms: BI 695501 prefilled syringe
Drug: BI 695501 autoinjector
  Arms: BI 695501 autoinjector

SUMMARY:
To investigate and compare the pharmacokinetics, safety and tolerability of BI 695501 administered subcutaneously via prefilled syringe or autoinjector

ELIGIBILITY:
Inclusion criteria:

* Healthy male, non-athletic* Caucasian subjects according to the investigator's assessment, based on a complete medical history including a physical examination, vital signs (blood pressure [BP], pulse rate [PR]), 12-lead ECG, and clinical laboratory tests.
* Age between 18 and 65 years (inclusive)
* BMI of 18 to 30 kg/m2 (inclusive)
* BMI 18 to <20, or
* BMI 20 to <25, or
* BMI 25 to <=30
* Signed and dated written informed consent prior to admission to the trial in accordance with Good Clinical Practice (GCP) and local legislation.
* Subjects agree to use an acceptable method of contraception during the trial and for 6 month after the dose of trial drug.

  * Non-athletic defined as person performing no more than one hour of exercise per week

Exclusion criteria:

* Any finding in the medical examination (including BP, PR or ECG) that deviates from normal and judged as clinically relevant by the investigator.
* Any evidence of a concomitant disease judged as clinically relevant by the investigator including gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders or diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts.
* Chronic or relevant acute infections.
* Positive result for HIV, HBV, and hepatitis C (Hep C) at screening.
* History of relevant allergy or hypersensitivity including allergy to the trial medication, its excipients or device materials (e.g. natural rubber or latex).
* Intake of drugs with a long half-life (more than 24 hours) within 30 days or less than 5 half-lives of the respective drug prior to administration of trial medication.
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial.
* Previous exposure to a biologic drug.
* Intake of an investigational drug in another trial within 2 months prior to intake of trial medication in this trial or intake of an investigational drug during the course of this trial.
* Smoker (more than 10 cigarettes or 3 cigars or 3 pipes per day).
* Inability to refrain from smoking during days of confinement at the trial site.
* Alcohol abuse (consumption of more than 4 units/day).
* Unwillingness/inability to refrain from intake of alcoholic beverages from 48 hours prior to the trial medication administration and until Day 14 post trial medication administration; and/or to limit alcohol intake to a maximum of 3 units per day until e.o.t.
* Drug abuse or positive drug screening.
* Blood donation of more than 100 mL within 30 days prior to administration of trial medication or intended donation during the trial.
* Intention to perform excessive physical activities within 1 week prior to administration of trial medication or contact sport during the entire trial and unwilling to avoid vigorous exercise for 14 days post dosing.
* Inability to comply with dietary regimen of trial site.
* Any out-of-range laboratory values considered clinically significant by the investigator; subjects with creatine kinase (CK) values 2 times the upper limit of normal (ULN) at Day -1 are excluded from participation.
* Subject is assessed as unsuitable for inclusion by the investigator, for instance, because he is considered not able to understand and comply with trial requirements, or has a condition that would not allow safe participation in the trial.
* Subjects with any immunological disorders or auto-immune disorders, (e.g., RA, lupus erythematosus, scleroderma, etc.).
* Subject has received a live vaccine within 12 weeks prior to enrolling in the trial.
* History of TB or positive finding in IGRA.
* Evidence of skin irritation or infection at the planned injection place.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2015-10-28 (Actual); Primary Completion 2016-09-07 (Actual); Study Completion 2016-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- SGS Belgium NV Research Unit Stuivenberg, Antwerp, Belgium

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was randomized, single-dose, parallel-arm, open-label Phase I trial with healthy male subjects.
Groups:
- BI 695501 Autoinjector (AI): Subject received single dose of 40 milligram (mg)/ 0.8 milliliters (mL) BI 695501 solution for injection in auto injector via subcutaneous injection followed by a 43-day observation period and up to 70 days safety follow-up period. (Test Product)
- BI 695501 Pre-filled Syringe (PFS): Subject received single dose of 40 milligram (mg)/ 0.8 milliliters (mL) BI 695501 solution for injection in pre-filled syringe via subcutaneous injection followed by a 43-day observation period and up to 70 days safety follow-up period. (Reference Product)
Period: Overall Study
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS)
Started | 35 | 36
Completed | 35 | 36
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects randomized set (RND): The RND consisted of all subjects in the subjects enrolled set (all subjects who provided informed consent for this trial.) who were randomized to trial medication. For analyses and displays based on RND, subjects were classified according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS) | Total
Number analyzed (Participants) | 35 | 36 | 71
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (13.77) | 40.1 (13.32) | 39.7 (13.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 35 | 36 | 71

OUTCOME MEASURES:

1. Primary Outcome: Maximum Measured Concentration of BI 695501 in Plasma (Cmax)
Description: Maximum measured concentration of BI 695501 in plasma (Cmax). The rate and extent of absorption of BI 695501 by assessment of maximum plasma concentration following administration via AI or via PFS of a single dose of 40 mg BI 695501. During analysis, it was realized that the PK sample on Day 43 had originally been mistakenly associated with a 1032 h time point, rather than with 1008 h. However, PK parameters are calculated using actual values so this did not impact the analysis results.
Time Frame: PK plasma samples were taken at: 1 hour (h) before drug administration and 1h, 4h, 8h,12h, 24h, 48h, 60h, 72h, 84h, 96h, 108h, 120h, 132h, 144h, 168h, 216h, 336h, 504h, 672h, 840h, 1008h after drug administration.
Population: Pharmacokinetic analysis set (PKS): The PKS consisted of all randomized subjects who received the single dose of trial medication, had at least one evaluable primary pharmacokinetic parameter, and were without important protocol deviations or violations thought to significantly affect the pharmacokinetics of BI 695501.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Micro-gram (µg) per milliliter (mL)
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS)
Number analyzed (Participants) | 35 | 36
Micro-gram (µg) per milliliter (mL) | 3.79 (27.4) | 3.48 (51.0)
Statistical Analysis 1: Comparison: BI 695501 Autoinjector (AI) vs BI 695501 Pre-filled Syringe (PFS); Analysis of variance (ANOVA) model on the log scale was used including treatment and body mass index (BMI) group as fixed effects; Test type: Superiority or Other; ANOVA; Ratio of adjusted geometric means (%) = 110.19, 90% CI 2-sided [96.80 to 125.44], Standard Deviation 33.603 — Relative bioavailability was estimated by the ratio (AI/PFS) of the adjusted geometric means (gMean). Standard deviation is actually inter-individual geometric coefficient of variation (%)

2. Primary Outcome: Area Under the Concentration-time Curve of the BI 695501 in Plasma Over the Time Interval From 0 to 1032 Hours After Dose (AUC0-1032)
Description: Area under the concentration-time curve of the BI 695501 in plasma over the time interval from 0 to 1032 hours after dose (AUC0-1032). The rate and extent of absorption of BI 695501 by assessment of AUC0-1032 following administration via AI or via PFS of a single dose of 40 mg BI 695501. During analysis, it was realized that the PK sample on Day 43 had originally been mistakenly associated with a 1032 h time point, rather than with 1008 h. However, PK parameters are calculated using actual values so this did not impact the analysis results.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS)
Number analyzed (Participants) | 35 | 35
μg*h/mL | 1810 (47.5) | 1840 (47.1)
Statistical Analysis 1: Comparison: BI 695501 Autoinjector (AI) vs BI 695501 Pre-filled Syringe (PFS); Analysis of variance (ANOVA) model on the log scale was used including treatment and BMI group as fixed effects; Test type: Superiority or Other; ANOVA; Ratio of adjusted geometric means (%) = 100.14, 90% CI 2-sided [85.15 to 117.76], Standard Deviation 42.354 — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Area Under the Concentration-time Curve of the BI 695501 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-infinity)
Description: Area under the concentration-time curve of the BI 695501 in plasma over the time interval from 0 extrapolated to infinity (AUC0-infinity) based on observed concentration at time of last measurable concentration. The rate and extent of absorption of BI 695501 by assessment of (AUC0-∞) following administration via AI or via PFS of a single dose of 40 mg BI 695501. During analysis, it was realized that the PK sample on Day 43 had originally been mistakenly associated with a 1032 h time point, rather than with 1008 h. However, PK parameters are calculated using actual values so this did not impact the analysis results.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg*h/mL
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS)
Number analyzed (Participants) | 35 | 35
μg*h/mL | 2080 (58.2) | 2110 (58.0)
Statistical Analysis 1: Comparison: BI 695501 Autoinjector (AI) vs BI 695501 Pre-filled Syringe (PFS); Analysis of variance (ANOVA) model on the log scale was used including treatment and BMI group as fixed effects; Test type: Superiority or Other; ANOVA; Ratio of adjusted geometric means (%) = 100.22, 90% CI 2-sided [82.13 to 122.29], Standard Deviation 53.137 — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Number of Subjects With Drug-related Adverse Events (AEs)
Description: Number of subjects with drug-related Adverse Events (AEs). Any event with an onset after the administration of the trial medication up to a period of 70 days was defined as a treatment-emergent AE (TEAE). A treatment-related AE was defined as any TEAE assessed by the investigator as related to the trial medication.
Time Frame: From the first drug administration until 43 days observation period after drug administration and up to 70 days safety follow up period
Population: Safety analysis set (SAF): The SAF consisted of all subjects in the enrolled set who received at least one dose of trial medication and subjects were classified according to treatment received.
Measure: Number; unit: Number of Subjects
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS)
Number analyzed (Participants) | 35 | 36
Number of Subjects | 20 | 16

ADVERSE EVENTS:
Time Frame: From the first drug administration until 43 days observation period after drug administration and up to 70 days safety follow up period
Description: Regular investigator assessment at study visits. The safety analysis set was used which consisted of all subjects who provided informed consent and who received at least one dose of trial medication.
Arm/Group | BI 695501 Autoinjector (AI) | BI 695501 Pre-filled Syringe (PFS)
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 28/35 | 23/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 Autoinjector (AI) (N=35) | BI 695501 Pre-filled Syringe (PFS) (N=36)
Fatigue (General disorders) | 1 | 2
Influenza like illness (General disorders) | 0 | 2
Injection site erythema (General disorders) | 18 | 13
Injection site induration (General disorders) | 4 | 1
Injection site pain (General disorders) | 3 | 0
Injection site pruritus (General disorders) | 1 | 2
Injection site swelling (General disorders) | 7 | 3
Nasopharyngitis (Infections and infestations) | 8 | 2
Contusion (Injury, poisoning and procedural complications) | 3 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Headache (Nervous system disorders) | 4 | 6
Paraesthesia (Nervous system disorders) | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.